CLINICAL TRIAL: NCT05881018
Title: Investigating the Effects of Diet and Physical Activity on Esport Performance
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Beneo-Institute (Industry)
Collaborators: German Sport University, Cologne (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: ES01
Record Dates: First submitted 2023-04-12; First posted 2023-05-30 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2023-05

CONDITIONS: Sports Physical Therapy; Dietary Habits; Diet, Healthy
MeSH Terms: conditions — Feeding Behavior | interventions — Exercise

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Low glycaemic index (Experimental)
  Interventions: Dietary Supplement: Low glycaemic index
- Low glycaemic index with physical activity units (Experimental)
  Interventions: Dietary Supplement: Low glycaemic index; Behavioral: Physical activity
- High glycaemic index (Experimental)
  Interventions: Dietary Supplement: High glycaemic index
- High glycaemic index with physical activity units (Experimental)
  Interventions: Dietary Supplement: High glycaemic index; Behavioral: Physical activity

INTERVENTIONS:
Dietary Supplement: Low glycaemic index — Diet will be supplemented with a drink containing a low glycaemic index carbohydrate
  Arms: Low glycaemic index; Low glycaemic index with physical activity units
Dietary Supplement: High glycaemic index — Diet will be supplemented with a drink containing a high glycaemic index carbohydrate
  Arms: High glycaemic index; High glycaemic index with physical activity units
Behavioral: Physical activity — Participants will include physical activity units
  Arms: High glycaemic index with physical activity units; Low glycaemic index with physical activity units

SUMMARY:
A randomized, counterbalanced intervention study in esport players.

DETAILED DESCRIPTION:
The study will test whether i) the consumption of two different carbohydrate drinks and ii) the performance of regular high-intensity interval training will impact esport performance and metabolic profile.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent obtained
* Male or female aged 18-45 years
* Healthy
* Participants have to be part of an esport association and/or regularly participate in tournaments

Exclusion Criteria:

* diabetes mellitus type 1 or 2 (T1DM or T2DM)
* medication which impacts glucose metabolism or visual perception
* health issues like cardiovascular diseases, severe orthopaedic conditions or neurological impairments
* food allergies or intolerances, e.g. fructose malabsorption

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 54 (Actual)
Dates: Start 2023-07-01 (Actual); Primary Completion 2023-12-01 (Actual); Study Completion 2023-12-01 (Actual)

PRIMARY OUTCOMES:
Change in esport performance (test battery) | 4 weeks
  Reaction time will be measured using an esport test battery

SECONDARY OUTCOMES:
Glucose response (continuous glucose monitor): 3h iAUC | 4 weeks
  The 3h incremental area under the curve (iAUC) will be used to assess glycemic response to the drink. Unit: mg/dL
Glycaemic variability (continuous glucose monitor): 24h MAGE | 4 weeks
  The mean amplitude of glycemic excursion during 24h will be assessed as an indicator for glycemic variability. Unit: mg/dL

CONTACTS AND LOCATIONS:
Locations (1):
- German Sports University Cologne, Cologne, Germany

IPD SHARING:
Plan to Share IPD: No